CLINICAL TRIAL: NCT05776784
Title: Status of Dental Care Practices in Patients With Hereditary Angioedema
Acronym: PRADA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC22.0357
Record Dates: First submitted 2023-02-24; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Angio Edema Hereditary
Keywords: prophylaxis; dental procedures
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — Dental Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: dental procedure — questionnaire for patient with dental procedure

SUMMARY:
Hereditary angioedema (HAE) is a rare genetic disease, it can occur at any age and evolves in flare-ups. These are subcutaneous or submucosal edemas responsible for tightness and pain. All areas can be reached. In addition, all their life, patients have an unpredictable risk of death from asphyxiating angioedema (25% mortality in the absence of specific treatment).

Surgical procedures, endoscopies and dental procedures can trigger laryngeal AE. Thus, the national reference center for angioedema (CREAK) and the latest international consensus1 recommend that all these procedures be preceded by short-term prophylaxis. The reference treatment is the C1 inhibitor 2 concentrate. But to date, there is no prospective study that has demonstrated the effectiveness of this short-term prophylaxis before dental treatment. Only a retrospective study has shown that its implementation made it possible to reduce the risk of crisis by 42% after tooth extraction 3 and that the risk of crisis was greatest within 8 hours following tooth extraction.

The C1 inhibitor concentrate must be administered IVL by a nurse within 6 hours before the procedure and therefore implies, in addition to its high cost (1500 €), an organizational burden for the patient who must plan for the passage of an IDE, the availability of the product and this sometimes for a simple dental treatment.

These constraints have two consequences for dental care: patients avoid going to the dentist to the detriment of their dental health or do not take prophylaxis with the risk of a fatal attack.

ELIGIBILITY:
Inclusion Criteria:

* Patient with HAE with or without C1 Inhibitor deficiency
* Patient over 18 years old

Exclusion Criteria:

* Patient opposed to the use of their data or refusing to answer the questionnaire
* Adult patients protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with HAE with or without C1 Inhibitor deficiency
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
the attitude of HAE patients towards dental care | 30 minutes
  Proportion of patients canceling or delaying dental care due to apprehension of a crisis or difficulties in scheduling short-term prophylaxis

SECONDARY OUTCOMES:
Description of crises after dental care | 30 minutes
  Proportion of patients with an attack within 48 hours after treatment, severity and location, Short-term prophylaxis used, Long-term prophylaxis used, Types of angioedema

CONTACTS AND LOCATIONS:
Locations (1):
- chu grenoble alpes CREAK, Grenoble, France

IPD SHARING:
Plan to Share IPD: No